CLINICAL TRIAL: NCT00826059
Title: A Multicenter, Randomized, Double Blind, Sham Control, Parallel Arm Trial to Assess Effectiveness and Safety of the Ischemic Stroke System ISS, as an Adjunct to Standard of Care in Subjects With Acute Ischemic Stroke
Brief Title: Implant for Augmentation of Cerebral Blood Flow Trial, Effectiveness and Safety in a 24 Hour Window
Acronym: ImpACT-24B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLP1000500
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; randomized clinical trial; effectiveness; safety
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Stimulation (Active Comparator): Implantation/ISS Stimulation during 5 consecutive days & Standard of Care (SoC).
  Day 1: First stimulation initiated within 24 hours from stroke onset, following implantation completion. All subjects will be treated according to SoC for treatment of Acute Ischemic Stroke.
  Day 2-4: ISS Stimulation treatment sessions repeated daily. Each treatment will be initiated within 18-26 hours from the preceding treatment.
  Day 5: Following completion of the last ISS Stimulation treatment session, imaging performed for assessing Injectable Neuro Stimulator (INS) positioning and/or lesion. Implant removal procedure will then be performed. Subsequently, patients will be evaluated for safety and effectiveness.
  Subjects will continue with SoC as needed and discharged from the hospital based on the judgment of the study investigator.
  Interventions: Device: Active Sphenopalatine Ganglion (SPG) Stimulation
- Sham Stimulation (Sham Comparator): Sham Implantation and Sham Stimulation during 5 consecutive days & Standard of Care (SoC).
  Day 1: First Sham stimulation initiated within 24 hours from stroke onset, following Sham implantation procedure. All subjects will be treated according to SoC for treatment of Acute Ischemic Stroke.
  Day 2-4: Sham Stimulation sessions repeated daily. Each Sham Stimulation will be initiated within 18-26 hours from the preceding treatment.
  Day 5: Following completion of the last Sham Stimulation session, imaging performed for lesion assessment. Sham Implant removal will then be performed. Subsequently, patients will be evaluated for safety and effectiveness.
  Subjects will continue with SoC as needed and discharged from the hospital based on the judgment of the study investigator.
  Interventions: Device: Sham Sphenopalatine Ganglion (SPG) Stimulation

INTERVENTIONS:
Device: Active Sphenopalatine Ganglion (SPG) Stimulation — SPG stimulation and standard of care. During all study periods, patients will receive Standard of Care in accordance to the general management of ischemic stroke and secondary prevention, following the guidelines of the American Heart Association/American Stroke Association and of the European Stroke Organization (ESO), including the use of antiplatelets, management of secondary stroke, dyslipidemia, hypertension, diabetes and counseling regarding smoking cessation. Off-label uses of drugs and devices should not occur during any of the study periods.
  Other Names: Standard of Care
  Arms: Active Stimulation
Device: Sham Sphenopalatine Ganglion (SPG) Stimulation — Sham SPG stimulation and standard of care. During all study periods, patients will receive Standard of Care in accordance to the general management of ischemic stroke and secondary prevention, following the guidelines of the American Heart Association/American Stroke Association and of the European Stroke Organization (ESO), including the use of antiplatelets, management of secondary stroke, dyslipidemia, hypertension, diabetes and counseling regarding smoking cessation. Off-label uses of drugs and devices should not occur during any of the study periods.
  Other Names: Standard of Care
  Arms: Sham Stimulation

SUMMARY:
The primary objective of the study is to assess the safety and effectiveness of SPG stimulation with the ISS in patients with an acute ischemic stroke in the anterior circulation initiated within 24 hours from stroke onset.

DETAILED DESCRIPTION:
A multi-center, multinational, randomized, blinded, sham control, adjunctive to Standard of Care, parallel arm study and will include ongoing Data Safety and Monitoring Board (DSMB) review of accumulated safety data.

Screening:

Since the treatment should be initiated within 24 hours from stroke onset, the screening window is limited and all procedures should be performed within this window.Subjects with Acute Ischemic Stroke will be screened upon arrival to the hospital. Since the treatment should be initiated between 8 and 24 hours from stroke onset, the screening window is limited and all procedures should be performed as soon as possible. All screened patients will be identified by patient number and will sign the informed consent prior to any study procedure initiation.

Period 1: Day 1-5

Day 1- Eligible subjects will be randomized to:

* Group 1: Implantation and ISS Stimulation during five consecutive days & Standard of Care
* Group 2: Sham Implantation and Sham Stimulation during five consecutive days & Standard of Care Subjects will be transferred to the implantation procedure facility and the implantation/sham implantation will be performed by a trained physician.

After implantation, active/sham stimulation will be administered in daily 4-hour sessions, beginning immediately following the placement procedure and continuing for 5 consecutive days.

Day 5 / Day of Discharge. Following the last ISS /Sham Stimulation, explantation will be performed and the patients will be evaluated for safety and effectiveness.

Subjects will continue with Standard of Care as needed and will be released from the hospital upon investigator's judgment.

Period 2: Day of Discharge - 89±7 days During this period both groups (ISS Stimulation and Sham Control) will be treated according to Standard of Care either at the hospital, rehabilitation center or at home.

Scheduled visits will be performed on day 30±7 and day 60 ±7, which will include safety and effectiveness assessments.

Final Visit Day 90±7 days: The final visit will be performed at the study site and will include safety and effectiveness evaluations.

Patients will be contacted by study personnel via telephone on Day 180±7 and on Day 360±7 in order to assess their quality of life status.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Between 40 years and 80 years for male and 85 for female subjects
2. Clinical diagnosis of an acute ischemic stroke in the Carotid, Middle or Anterior Cerebral Artery territories
3. Imaging findings demonstrating signs of ischemia in the anterior circulation, consistent with the clinical diagnosis
4. Baseline NIHSS ≥ 7 and ≤ 18 within 2 hours prior to implantation.
5. Ability to initiate treatment within 8- 24 hours from stroke onset
6. Signed informed consent from patient him/herself or legally authorized representative if applicable

Exclusion Criteria:

1. Intracranial hemorrhage or hemorrhagic transformation
2. Massive stroke
3. Acute ischemic stroke in the posterior circulation
4. Minor stroke
5. Treated with IV-tPA (intravenous tissue Plasminogen Activator) ,IA-tPA (intra-arterial tissue Plasminogen Activator) or neurothrombectomy devices for the current stroke
6. Previous stroke in the last 6 months or pre-existing disability
7. Patients with bleeding propensity or any condition in the oral cavity that prevents implantation
8. Clinical signs and symptoms or imaging evidence of bilateral stroke.
9. Treated with IV-tPA ,IA-tPA or neurothrombectomy devices for the current stroke.
10. Known cerebral arteriovenous malformation, cerebral aneurysm.
11. Clinical suspicion of septic embolus.
12. Uncontrolled hypertension (systolic >185 mmHg and/or diastolic >110 mmHg)
13. Serious systemic infection.
14. Women known to be pregnant or having a positive or indeterminate pregnancy test.
15. Patients with other implanted neural stimulator/ electronic devices (pacemakers).
16. Life expectancy < 1 year from causes other than stroke.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1078 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Sliding Dichotomy modified Rankin Scale (mRS) at 3 months | 90 days±7 days
  The primary efficacy endpoint is improvement beyond expectations on the modified Rankin Scale at 3 months (sliding dichotomy), assessed in primary populations of:
  1. modified intention to treat (mITT)
  2. confirmed cortical involvement (CCI), defined as baseline NIHSS ≥ 10 and signs of cortical involvement in baseline imaging (at least one of the following ASPECT regions: M1-M6, Insular Cortex) Type I Error is controlled at an overall level of 0.05 (two-sided) using the Hochberg method.

OTHER OUTCOMES:
Subgroup analysis | 90 days±7 days
  Primary parameters subgroup analysis by: NIHSS strata, lesion size, time from stroke onset strata, gender, age strata, Diabetes (Y/N), Atrial Fibrillation AFIB (Y/N) and side
Additional clinical efficacy outcome: SIS-16 | 90 days±7 days
  Stroke-related quality of life at 3 months according to the Stroke Impact Scale-16 (SIS-16)
Additional clinical efficacy outcome: Dichotomy 0-2 mRS at 3 months | 90 days±7 days
  Functional independence at 3 months (modified Rankin Scale 0-2)
Additional clinical efficacy outcome: Dichotomy 0-3 mRS at 3 months | 90 days±7 days
  Up to moderate disability but ambulatory at 3 months (modified Rankin Scale 0-3)
Safety outcome: Serious Adverse Event (SAE) | 90 days±7 days
  All Serious Adverse Events (SAEs)
Safety outcome: Serious Adverse Event (SAE) - Implantation | 90 days±7 days
  SAEs related to implant placement or removal
Safety outcome: Serious Adverse Event (SAE) - Stimulation | 90 days±7 days
  SAEs related to stimulation
Safety outcome: Neurological Deterioration | 10 days
  An increase of 4 or more points on the NIHSS related to any neurological event within the first 10 days after stroke onset
Safety outcome: Mortality | 90 days±7 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shay, Study Director — BrainsGate
Locations (73):
- United States (7):
  - Intercoastal Medical Group, Sarasota, Florida
  - Central DuPage Hospital, Winfield, Illinois
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - University of Toledo Medical Center- Campus 1, Toledo, Ohio
  - University of Toledo Medical Center- Campus 2, Toledo, Ohio
  - Palmetto Health Richland, Columbia, South Carolina
  - Erlanger Stroke Center, Chattanooga, Tennessee
- Canada (2):
  - Foothills Medical Centre/University of Calgary, Department of Clinical Neurosciences, Calgary
  - Department of Medicine, Stroke Program, University of Alberta Hospital, Edmonton
- Czechia (3):
  - University Hospital of Ostrava, Ostrava Poruba, Poruba
  - General University Hospital, Prague
  - Vitkovicka nemocnice a.s. Ostrava Vitkovice, Vítkovice
- Aarhus University Hospital, Aarhus, Denmark
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- France (5):
  - Hospital de la Cavale Blanche, Brest
  - Hospital Nord Laennec, Nantes
  - Hospital Saint Roch, Nice
  - Hopital Lariboisiere, Paris
  - Hospital Pontchaillou, Rennes
- Georgia (7):
  - Unimed Adjara Batumi Referral Hospital, Batumi
  - Kutaisi Referral Hospital, Kutaisi
  - Rustavi Central Hospital, Rustavi
  - Emergency Neurology Clinic Neurology Ltd., Tbilisi
  - First University Clinic, Tbilisi
  - High Technology Medical Center University Clinic LTD., Tbilisi
  - Zugdidi Referral Hospital, Zugdidi
- Germany (9):
  - Altenburg Clinic of Neurology, Altenburg
  - Bad Neustadt Neurological Clinic, Bad Neustadt an der Saale
  - Center for Stroke Research at Charite University of Berlin, Berlin
  - Erlangen University Clinic, Erlangen
  - Essen University Clinic, Essen
  - Heidelberg University Clinic, Heidelberg
  - Leipzig University Clinic, Leipzig
  - Technical University Munich, Munich
  - Schwarzwald-Baar Clinic, Villingen-Schwenningen
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (2):
  - Hospital Sant'Andrea delle Fratte, Perugia
  - Policlinico Umberto I, Roma
- University Clinic for Neurology, Skopje, North Macedonia
- Poland (6):
  - Bialystok University Hospital, Bialystok
  - Konske Hospital, Gmina Końskie
  - University Hospital in Krakow, Krakow
  - Sandomierz Hospital, Sandomierz
  - Torun Hospital, Torun
  - Institute of Psychiatry and Neurology, Warsaw
- Portugal (4):
  - Hospital Fernando Fonseca, Amadora
  - Hospital de Santo Antonio, Porto
  - Unidade de AVC Centro Hospitalar São João, Porto
  - Centro Hospitalar de Douro e Vouga, EPE - Hospital de São Sebastião, Santa Maria
- Serbia (3):
  - Special Hospital for Cerebrovascular Disease Sveti Sava, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
  - Clinical Hospital Center Zemun, Zemun
- Slovakia (2):
  - Neurologické Oddelenie, Nemocnica s Poliklinikou Spišská, Nová Ves
  - Neurologické Oddelenie FN Trnava, Fakultná Nemocnica, Trnava
- Spain (11):
  - Hospitalario Universitario de Albacete, Albacete
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Gregorio Maranon, Madrid
  - Ramon Y Cajal, Madrid
  - Hospital Universitario Son Dureta, Palma de Mallorca
  - Complejo Hospitalarion Univiersitario de Santiago, Santiago de Compostela
  - Valladolid - Hospital Clinico, Valladolid
- Lviv National Medical University, Lviv, Ukraine

REFERENCES:
- [Derived] Bornstein NM, Saver JL, Diener HC, Gorelick PB, Shuaib A, Solberg Y, Thackeray L, Savic M, Janelidze T, Zarqua N, Yarnitsky D, Molina CA; ImpACT-24B investigators. An injectable implant to stimulate the sphenopalatine ganglion for treatment of acute ischaemic stroke up to 24 h from onset (ImpACT-24B): an international, randomised, double-blind, sham-controlled, pivotal trial. Lancet. 2019 Jul 20;394(10194):219-229. doi: 10.1016/S0140-6736(19)31192-4. Epub 2019 May 24. PMID 31133406